CLINICAL TRIAL: NCT07161518
Title: Characterizing Transcranial Focused Ultrasound Neuromodulation During Sedation
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Boris D. Heifets, Associate Professor of Anesthesiology, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 79882
Record Dates: First submitted 2025-08-14; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Active then Sham (Experimental): Active (focused) ultrasound followed by washout of 5 days or greater, followed by sham (unfocused) ultrasound
  Interventions: Device: Low-intensity transcranial ultrasound; Drug: Propofol
- Sham then Active (Experimental): Sham (unfocused) ultrasound followed by washout of 5 days or greater, followed by active (focused) ultrasound
  Interventions: Device: Low-intensity transcranial ultrasound; Drug: Propofol

INTERVENTIONS:
Device: Low-intensity transcranial ultrasound — Active (focused) ultrasound
Device: Low-intensity transcranial ultrasound — Sham (unfocused) ultrasound
Drug: Propofol — Intravenous propofol administration

SUMMARY:
The goal of this clinical trial is to learn if focused ultrasound delivered to the brain influences the effects of the anesthetic medication propofol. It will also learn about the safety and feasibility of using ultrasound and anesthesia together to influence the brain. The main questions it aims to answer are:

* Does focused ultrasound delivered to the brain influence the effects or the strength of propofol?
* Does propofol anesthesia influence the effects of ultrasound delivered to the brain?

Researchers will compare focused ultrasound with sham ultrasound (similar technology but not targeted to a brain region) and administer propofol anesthesia, while measuring signals from the brain and behaviors of participants.

Participants will:

* Obtain one non-contrast MRI scan of the brain
* Receive two separate sessions of ultrasound to the brain (one focused and one sham)
* Undergo two separate sessions of propofol anesthesia in a laboratory

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 65 years of age, inclusive, at time of screening.
2. Body mass index between 17-35 kg/m2.
3. Able to read, understand, and provide written, dated informed consent prior to screening. Participants will be deemed likely to comply with study protocol and communicate with study personnel about adverse events and other clinically important information.
4. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following specific criteria:

   1. Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized (status post hysterectomy, bilateral tubal ligation), or is post-menopausal with her last menses at least one year prior to screening); or
   2. Childbearing potential, and meets the following criteria:

   (i) Negative urinary pregnancy test at screening, confirmed by a negative urinary pregnancy test at enrollment prior to receiving study treatment.

(ii) Willing and able to continuously use one of the following methods of birth control during the course of the study, defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly: implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence. The form of birth control will be documented at screening and baseline.

Exclusion Criteria:

1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
2. Female that is pregnant or breastfeeding.
3. Female with a positive pregnancy test at screening or baseline.
4. Current diagnosis of Axis I or II disorders other than Major Depressive Disorders, Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Social Phobia, Specific Phobia, Obsessive-Compulsive Disorder, Post-Traumatic Stress Disorder, Somatization Disorder, Pain Disorder, Sexual and Gender Identity Disorders, Insomnia, Adjustment Disorders, Tic Disorders, and Neurodevelopmental Disorders.
5. Current diagnosis of Axis I disorders other than Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, Specific Phobia, or Bipolar II Disorder (unless one of these is comorbid and clinically unstable, and/or the focus of the participant's treatment for the past six months or more) History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes.
6. Any neurological disorder including:

   1. Dementia, delirium, amnestic, or any other cognitive disorder
   2. Lifetime history of surgical procedures involving the brain or meninges
   3. Encephalitis, meningitis, degenerative central nervous system disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, developmental delay
   4. Any other disease/procedure/accident/intervention associated with significant injury to or malfunction of the central nervous system (CNS),
   5. History of significant head trauma resulting in cognitive impairment within the past two years.
7. Any cardiovascular disorder including:

   1. Uncontrolled hypertension
   2. Congestive heart failure NYHA Criteria >Stage 2
   3. Atrial fibrillation or resting heart rate <50 or >105 beats per minute at screening
   4. Clinicially significant uncontrolled arrhythmia
   5. QTcF (Fridericia-corrected) >= 450 msec at screening
   6. Any cardiovascular disorder that would merit categorization of patient as ASA Class 3 or higher
8. Any pulmonary/respiratory disorder including:

   1. Formally diagnosed obstructive sleep apnea (OSA) that is moderate and not treated with a CPAP machine; or formally diagnosed OSA that is severe, regardless of treatment
   2. Undiagnosed OSA with a STOPBANG score of 5 or higher
   3. History of difficult airway in surgical setting
   4. Any pulmonary/respiratory disorder that would merit categorization of patient as ASA Class 3 or higher
9. Clinically significant liver disease, determined by LFTs within the past 6 months
10. Clinically significant kidney disease determined by creatinine / GFR within the past 6 months
11. Symptomatic gastroesophageal reflux disease, hiatal hernia, taking medications causing delayed gastric emptying, or any other gastrointestinal disorder placing the patient at risk for aspiration or that would merit categorization of patient as ASA physical classification status of III or higher
12. Any endocrine disorder including:

    1. Uncontrolled diabetes mellitus, type 1 or 2
    2. Clinically significant hypothyroidism or hyperthyroidism which has not been stably treated for at least 6 months
    3. Any other endocrine disorder that would merit categorization of patient as ASA Class 3 or higher
13. Patients taking any of the following daily medications:

    1. Opioids including buprenorphine and methadone
    2. Naltrexone or other opioid antagonist
    3. Clonidine
14. Any other clinically significant abnormal laboratory result at the time of the screening exam that might affect safety, study participation or confound interpretation of study results
15. Any other clinically significant physical exam abnormality on the screening physical examination that might affect safety, study participation or confound interpretation of study results, including any condition that would merit categorization of patient as ASA Class 3 or higher
16. Participation in any clinical trial with an investigational drug or device that conflicts with this trial, within the past month or concurrent to study participation.
17. Abnormalities noted on anatomy mapping brain MRI as determined by radiologist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Electroencephalographic power spectral density | 3 hour period concurrent with delivery of propofol anesthesia
  Electroencephalographic (EEG) power will be computed using the multitaper spectrogram method applied to frontal, central, and posterior EEG leads and will be reported in the 0.5 Hz (delta) to 40 Hz (gamma) range inclusive of all bands therein (delta, theta, alpha, beta, gamma).

SECONDARY OUTCOMES:
Percent responsiveness to commands | 3 hours concurrent with delivery of propofol anesthesia
  Measured via electronically delivered commands and electronically monitored response button
Reaction time to verbal commands | 3 hours concurrent with delivery of propofol anesthesia
  Measured via electronically delivered verbal commands and electronically monitored response button
Reaction time in visual psychomotor vigilance test | Prior to delivery of propofol anesthesia, directly upon cessation of propofol anesthesia, and 15 minutes following cessation of propofol anesthesia
  Delivered via computer screen and button
Number of trials completed in 90-second digit symbol substitution test | Prior to delivery of propofol anesthesia, directly upon cessation of propofol anesthesia, and 15 minutes following cessation of propofol anesthesia
  Using a standardized protocol for the digit symbol substitution test delivered via computer screen and keyboard for participant responses
Pressure pain threshold | 15 minutes preceding the start of, and following cessation of, delivery of propofol anesthesia
  Measured via quantitative algometer testing on the trapezius muscle
Electroencephalographic power spectral density | 15 minutes preceding the start of, and following cessation of, delivery of propofol anesthesia
  Electroencephalographic (EEG) power will be computed using the multitaper spectrogram method applied to frontal, central, and posterior EEG leads and will be reported in the 0.5 Hz (delta) to 40 Hz (gamma) range inclusive of all bands therein (delta, theta, alpha, beta, gamma).

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No